CLINICAL TRIAL: NCT05943691
Title: High-dose Dexamethasone Plus Hetrombopag Versus High-dose Dexamethasone Alone as Frontline Treatment for Newly Diagnosed Adult Primary Immune Thrombocytopenia (ITP):A Prospective Multicenter Randomized Trial
Brief Title: High-dose Dexamethasone Plus Hetrombopag vs High-dose Dexamethasone Alone as Frontline Treatment for Newly Diagnosed Adult Primary Immune Thrombocytopenia: A Prospective, Multicenter, Randomized Trial
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Ming Hou, Professor and Director, Shandong University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ITP-Hetrombopag plus HD-DEX
Record Dates: First submitted 2023-07-05; First posted 2023-07-13 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: ITP - Immune Thrombocytopenia
Keywords: Hetrombopag, Dexamethasone
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — hetrombopag; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hetrombopag plus High-dose Dexamethasone (Experimental): Hetrombopag 5mg po qd; HD-DEX 40mg qd for 4 days
  Interventions: Drug: hetrombopag 5mg po qd; Drug: High-dose Dexamethasone
- High-dose Dexamethasone (Active Comparator): HD-DEX 40mg qd for 4 days
  Interventions: Drug: High-dose Dexamethasone

INTERVENTIONS:
Drug: hetrombopag 5mg po qd — hetrombopag 5mg po qd for 8 weeks, combining with dexamethasone 40 mg qd for 4 days
  Arms: Hetrombopag plus High-dose Dexamethasone
Drug: High-dose Dexamethasone — dexamethasone 40 mg qd for 4 days

SUMMARY:
The project was undertaking by Qilu Hospital of Shandong University in China. In order to report the efficacy and safety of Hetrombopag plus high-dose dexamethasone for the treatment of adults with newly-diagnosed primary immune thrombocytopenia (ITP).

DETAILED DESCRIPTION:
The investigators anticipate to undertaking a parallel group, randomised controlled trial of 100 ITP patients. One part of the participants are randomly selected to receive hetrombopag with starting dose 5mg po qd for 8 weeks（increase daily dose to a maximum of 7.5 mg/day if platelet count<50000 per μL following at least 2 weeks of treatment) combining with dexamethasone (given at a dose of 40 mg qd for 4 consecutive days). The others are selected to receive high-dose of dexamethasone alone. Patients who do not respond to dexamethasone may receive another cycle of high-dose dexamethasone therapy within 2 weeks. Platelet count, bleeding and other symptoms were evaluated before and after treatment. Adverse events are also recorded throughout the study. The purpose of this study is to report the efficacy and safety of Hetrombopag combining with high-dose dexamethasone therapy for the treatment of newly diagnosed ITP.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years
* Meet the diagnostic criteria for newly diagnosed immune thrombocytopenia (diagnosed within 3 month);
* platelet count <30*10^9/L, or < 50*10^9/L with bleeding manifestations, both;
* Willing and able to sign written informed consent

Exclusion Criteria:

* secondary thrombocytopenia or graded MF≥2 myelofbrosis based on the European Consensus Scale
* Previous history of treatment for ITP, except Platelet transfusion, ITP-directed Prednisone therapy no more than 2 weeks or TPO therapy no more than 1 week and stopped ≥1 week before randomization
* No response to TPO-RA or rhTPO
* HIV, hepatitis C or B virus infection
* pregnancy or lactation;
* arterial or venous thromboembolism within the 6 months before screening
* total bilirubinalanine, aminotransferase or aspartate transaminase>3×upper limit of normal (ULN), serum creatinine>1.5×ULN
* congestive heart failure (New York Heart Association [NYHA] class III/IV);
* neoplastic disease within the past 5 years;
* liver cirrhosis
* people who could not adhere to the protocol or were planning to have a surgical procedure in 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-09-15 (Estimated); Primary Completion 2024-07-10 (Estimated); Study Completion 2024-12-10 (Estimated)

PRIMARY OUTCOMES:
26 week sustained overall response to ITP treatments | 26-week after treatment started
  Complete response was defined as a platelet count of 100 000 per μL or higher and an absence of bleeding.
  Partial response was defined as a platelet count of 30000 per μL or higher,and at least a doubling of the baseline platelet count and an absence of bleeding.
  No response was defined as a platelet count of less than 30000 per μL, or less than two-times increase from baseline platelet count, or bleeding.

SECONDARY OUTCOMES:
28-day initial complete response to ITP treatment | 28 days after treatment started]
  Complete response was defined as a platelet count of 100 000 per μL or higher and an absence of bleeding.
  Partial response was defined as a platelet count of 30000 per μL or higher,and at least a doubling of the baseline platelet count and an absence of bleeding.
  No response was defined as a platelet count of less than 30000 per μL, or less than two-times increase from baseline platelet count, or bleeding.
28-day initial overall response to ITP treatment | 28 days after treatment started
  Complete response was defined as a platelet count of 100 000 per μL or higher and an absence of bleeding.
  Partial response was defined as a platelet count of 30000 per μL or higher,and at least a doubling of the baseline platelet count and an absence of bleeding.
  No response was defined as a platelet count of less than 30000 per μL, or less than two-times increase from baseline platelet count, or bleeding.
8-week complete response to ITP treatment | 8 weeks after treatment started
  Complete response was defined as a platelet count of 100 000 per μL or higher and an absence of bleeding.
  Partial response was defined as a platelet count of 30000 per μL or higher,and at least a doubling of the baseline platelet count and an absence of bleeding.
  No response was defined as a platelet count of less than 30000 per μL, or less than two-times increase from baseline platelet count, or bleeding.
8-week overall response to ITP treatment | 8 weeks after treatment started
  No response was defined as a platelet count of less than 30000 per μL, or less than two-times increase from baseline platelet count, or bleeding.
time to response | an average of 6 months
  the time from treatment initiation to achieve a complete response or a partial response
duration of response | through study completion, an average of one year
  the time from achievement of a complete response or a partial response to the loss of response
therapy associated adverse events | through study completion, an average of one year

CONTACTS AND LOCATIONS:
Locations (1):
- Shengli Oilfield Central Hospital, Dongying, Shandong, China